CLINICAL TRIAL: NCT03397810
Title: Effect of Radiotherapy on ATTR Cardiac Amyloidosis : a Proof of Concept Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philippe Meyer (Other)
Responsible Party: Sponsor-Investigator, Philippe Meyer, Principal Investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-00640
Record Dates: First submitted 2018-01-04; First posted 2018-01-12 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Amyloid Cardiomyopathy
Keywords: cardiac amyloidosis; radiotherapy
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Singe arm (Experimental): Subjects will receive a low dose radiotherapy focused to the heart
  Interventions: Radiation: low dose radiotherapy

INTERVENTIONS:
Radiation: low dose radiotherapy — 10 Gy in 5 fractions of 2 Gy on 5 consecutive days

SUMMARY:
Cardiac amyloidosis is responsible for significant morbidity associated with heart failure, and carries a poor prognosis. Currently there are very limited treatment options for this condition. Radiotherapy has been used successfully to treat amyloidosis elsewhere in the body, however has not been tried in cardiac amyloidosis. Therefore this study aims to assess the effect of radiotherapy on cardiac amyloidosis, to evaluate whether it can successfully reduce the burden of amyloid deposits in the myocardium as assessed by 18F-Amyloid PET.

DETAILED DESCRIPTION:
The intervention will involve administration of external beam radiotherapy (5 fractions of 2Gy) focused to the heart.

Measurements of effect will be assessed at 12 weeks by:

Amyloid PET Cardiac MRI with administration of gadolinium and ultrasound A blood venous sample (cardiac biomarkers) Quality of life assessments

ELIGIBILITY:
Inclusion Criteria:

* Age >65 y.o.
* Dyspnoea on exertion (NYHA II or more).
* Stable elevated cardiac enzymes (ultra sensitive Troponin T > 14 ng/L on consecutive sampling or BNP > 100pg/mL)
* A positive 99mTc-DPD cardiac scintigraphy (Grade 2 and 3) suggesting an ATTR or wt amyloidosis.
* Additional imaging also compatible with cardiac amyloidosis (cardiac ultrasound showing basal to apical longitudinal strain gradient and magnetic resonance imaging with elevated T1 value or extracellular volume).
* Compliance with the informed consent as attested by its signature.
* Positive baseline 18F-Florbetapir imaging, as assessed visually and quantitatively by a Tissue to Background Ratio > 1.45

Exclusion Criteria:

* Positive serum protein immunoelectrophoresis with monoclonal gammapathy.
* Previous external beam radiotherapy including the chest.
* Claustrophobia
* Presence of internal non-MR compatible devices
* Creatinine glomerular filtration rate < 30 ml/min
* Oncologic disease (excluding skin cancer) active or in remission from less than 5 years

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-03-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Assessment of the degree of amyloid | 12 weeks
  Assess intra-individual change in a quantitative measure of amyloid deposits on 18F-Amyloid (Standard Uptake Value ratio) SUVR between amyloid PET scans before and after low dose RT

SECONDARY OUTCOMES:
Safety and adverse event associated with cardiac low dose RT | 6 months
  Assess the number of patients who report adverse events
Modification in echocardiographic global longitudinal strain | 6 months
  Assess intra-individual change in a quantitative measures
Modification in MRI extracellular volumes and T1 values | 12 weeks
  Assess intra-individual change in a quantitative measures
Modification in cardiac biomarker (ultrasensitive troponin T and BNP blood levels) features of cardiac amyloidosis | 6 months
  Assess intra-individual change in a quantitative measures
Modification of quality of life | 6 months
  The quality of life will be assessed by the SF-36 short form health survey quality of life scale

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided